CLINICAL TRIAL: NCT01429363
Title: Targeted Disc Decompression (TDD) for Contained Herniated Lumbar Discs. A Prospective Clinical Series
Brief Title: Targeted Disc Decompression (TDD) for Contained Herniated Lumbar Discs
Acronym: TDD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: NeuroTherm (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTC 760-220411
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Lumbar Spine Disc Herniation
Keywords: contained herniated lumbar discs; TDD; Case series; RCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Targeted disc decompression (Experimental)
  Interventions: Procedure: Targeted disc decompression

INTERVENTIONS:
Procedure: Targeted disc decompression — The Targeted disc catheter is connected to Neurotherm TDD unit and heating protocol is started.In this heating protocol temperature gradually increases from 65C to 90C during a time period of 12 minutes;

SUMMARY:
The prospective Clinical Series (CS) aims to prove the hypothesis that Targeted Disc Decompression (TDD) reduces the pain in patients suffering from radicular leg pain secondary to a contained focal disc protrusion (Lumboradicular Syndrome). Secondary objective will be to prove that the treatment Group will have less disability and better quality of life.

DETAILED DESCRIPTION:
The study will start with a prospective clinical series (CS) in which 20 patients after careful selection will be treated with TDD, followed by a standardized rehabilitation program. After the diagnosis Lumboradicular syndrome the patient will first receive an transforaminal epidural injection at the site and level of the herniated disc, proven on MRI. Two weeks after the epidural injection the patient is evaluated. When the response is negative (a decrease less than 2.5 points on the 10 points VAS scale) TDD can be performed. Patient outcome will be evaluated at 6 weeks, 3, 6, 12 and 24 months after the study intervention. End point of this study is 3 months after TDD treatment. A positive response is defined as a minimal decrease of 2.5 points on the 10 points VAS scale compared to the VAS score at baseline.

A positive response in at least seven patients and acceptable side-effects and complications will lead to the start of a RCT.

If the response is positive < 7 out of 20 patients, the decision to proceed with a RCT following the prospective CS is made after evaluation of the CS by a team of experts. The results from this prospective study will be published.

ELIGIBILITY:
Inclusion Criteria:

* Mono radicular leg pain for at least 6 weeks as a result from a lumbar contained herniated disc. Leg pain must be of greater impact then concomitant back-pain
* Failing conservative treatment; analgesics and/or physical therapy ( WHO 1-3). Failing means persisting pain leading to problems with daily activities.
* MRI: must be performed < 6 weeks before start treatment. On MRI signs of contained herniated disc, maximum 33% obliteration of the spinal channel. No signs of other significant spine pathology (see exclusion criteria).
* Negative response to a transforaminal epidural injection. Injection must be performed < 6 weeks before start treatment but least 2 weeks before start treatment
* Neurological investigation by neurologist. Symptoms should be clinical related to the disc herniation level.
* Age >18 and < 50 years
* Mean pain on visual analogue scale (VAS) >50 mm (0 -100)

Exclusion Criteria:

* Herniated disc with more then 33% obliteration of the spinal channel.
* Annulus rupture with sequestrated herniated disc.
* Pain on VAS below 50 mm
* Pain existing longer then one year
* Less then 50% preserved disc height
* Conflict with social security/insurance
* Major motor impairment as a result of the herniation, paresis gr 3 MRC or more
* Other degenerative causes of nerve root compression; ligament flavum or facet joint hypertrophy, degenerative spinal channel stenosis, loss of lumbar kyphosis, discopathy with signs of Schmorls' nodules and loss of nucleus pulposus signal. Other causes of radicular syndrome such as cancer, radiculitis or neural degeneration.
* Spinal instability (spondylolisthesis, spinal fracture or tumor)
* History of back surgery, chemonucleolysis or other intra discal procedures
* Coagulopathies or oral anti-coagula therapy
* Infection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Primary end point is pain after 3 months measured by the 10 point Jensen's visual analogy scale | 3 months after treatment
  Primary end point is pain after 3 months measured by the 10 point Jensen's visual analogy scale. Patient outcome will be evaluated at 6 weeks, 3, 6, 12 and 24 months by a Anesthesiologist and the research nurse - both blinded for the performed procedure.

SECONDARY OUTCOMES:
MPQ-DLV (second pain measurement) | Patient outcome will be evaluated at 6 weeks, 3, 6, 12 and 24
Quebec Back Pain Disability Scale (disability) | Patient outcome will be evaluated at 6 weeks, 3, 6, 12 and 24
Rand-36 (quality of live) | Patient outcome will be evaluated at 6 weeks, 3, 6, 12 and 24
7-point Likert scale (global perceived effect) | Patient outcome will be evaluated at 6 weeks, 3, 6, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: JW Kallewaard, Drs., Principal Investigator — Rijnsate Hospital
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Diakonessenhuis, Utrecht, Utrecht
  - Rijnland Ziekenhuis, Leiderdorp